CLINICAL TRIAL: NCT03115515
Title: Randomized, Prospective Trial Comparing the Safety and Efficacy of Empiric Levothyroxine (LT4) Dose Increase Versus Individualized LT4 Dose Increase in Hypothyroid Women During Pregnancy
Brief Title: Safety and Efficacy of Empiric Levothyroxine (LT4) Dose Increase Versus Individualized LT4 Dose Increase in Hypothyroid Women During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Shannon Sullivan, Principal Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-235
Record Dates: First submitted 2017-04-07; First posted 2017-04-14 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy Related; Thyroid
Keywords: Thyroid Stimulating Hormone
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjustment in number of doses of thyroid hormone per week (Experimental): Patients in this group will increase pre-pregnancy thyroid hormone dose by 2 doses/week (extra dose on Wednesday and Saturday). Further dose adjustment are made every 2-4 weeks based on serum TSH, as shown below:
  * TSH>10mIU/L, increase by 3 doses/week
  * TSH 5.0-9.9mIU/L, increase by 2 doses/week
  * TSH 2.0-4.9mIU/L, increase by 1 dose/week
  * TSH 0.4-1.9mIU/L, no change
  * TSH<0.4mIU/L, decrease by 1 dose/week
  * TSH<0.1mIU/L, decrease by 2 doses/week
  * Thyroid hormone dose will NOT be decreased due to TSH<0.4mIU/L during the 1st trimester unless patient also has elevated circulating T4 and/or T3 levels, indicate of true hyperthyroidism.
  Interventions: Drug: levothyroxine
- Adjustment in micrograms per day of thyroid hormone (Experimental): Patients in this group adjust thyroid hormone dose based on Visit 1 TSH and pre-pregnancy thyroid hormone dose. Further dose adjustments are made every 2-4 weeks based on serum TSH, as shown below:
  * TSH>10mIU/L, increase dose by 50mcg/day if dose <125mcg/day or increase by 75mcg/day if dose >125mcg
  * TSH 5.0-9.9mIU/L, increase dose by 25mcg/day if dose <125mcg/day or increase by 50mcg/day if dose >125mcg
  * TSH 2.0-4.9mIU/L, increase dose by 12.5mcg/day if dose <125mcg/day or increase by 25mcg/day if dose >125mcg
  * TSH 0.4-1.9mIU/L, no change
  * TSH<0.4mIU/L, decrease dose by 12.5mcg/day if dose <125mcg/day or decrease by 25mcg/day if dose >125mcg/day
  * TSH<0.1mIU/L, decrease dose by 25mcg/day if dose <125mcg/day or decrease by 50mcg/day if dose >125mcg/day
  * Thyroid hormone dose will NOT be decreased due to TSH<0.4mIU/L during the 1st trimester unless patient also has elevated circulating T4 and/or T3 levels, indicate of true hyperthyroidism.
  Interventions: Drug: levothyroxine

INTERVENTIONS:
Drug: levothyroxine — To compare two different methods of adjusting thyroid hormone replacement during pregnancy to maintain TSH within the normal reference range for pregnancy.
  Other Names: Synthroid; Levoxyl

SUMMARY:
In women who require thyroid hormone replacement medication, the investigators will compare 2 ways to adjust thyroid medication during pregnancy to determine superiority in maintaining optimal blood levels of thyroid hormone. Thyroid hormone requirements increase significantly in pregnancy and it is important that blood levels of thyroid hormone remain normal so the fetus, which cannot make its own thyroid hormone has enough for early prenatal development. This trial compares 2 methods for adjusting thyroid medicine during pregnancy in women with known thyroid disease. Pregnant women (age 18 to 45) who take thyroid medication will be randomized to either 1) a 2-dose per week increase in thyroid medicine once pregnancy is confirmed, followed by dose adjustments every 2-4 weeks, or 2) adjustments in thyroid medication every 2-4 weeks in micrograms per day based on results of blood tests. The investigators will compare thyroid hormone levels throughout pregnancy between the groups of mothers to determine which method is superior in meeting the increased thyroid hormone requirements during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Female between ages of 18-45 who takes thyroid hormone replacement medicine AND pregnant or plan to become pregnant in the near future.

Exclusion Criteria:

* Males
* Younger than 18 or older than 45 years old
* More than 10 weeks pregnant at enrollment
* Iodine deficient
* Pregnant with more than one baby (i.e., twins, triplets, etc.)
* NOT taking thyroid hormone medicine before becoming pregnant
* Levels of thyroid hormone in blood have been too low or too high in the past 6 months
* Treated with radioactive iodine in the past year.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
% of TSH values within trimester-specific goal range per patient from study enrollment to delivery | TSH will be assessed every 2 weeks from enrollment to 28 weeks gestation and then every 4 weeks from 29 weeks to delivery
  % of TSH values within trimester-specific goal range according to study group

SECONDARY OUTCOMES:
Mean number of LT4 dose adjustment | Dose adjustments will be assessed every 2 weeks from enrollment to 28 weeks gestation and then every 4 weeks from 29 weeks to delivery
  Mean number of LT4 dose adjustments needed per patient in each group
Mean number of LT4 dose adjustments by hypothyroidism etiology | Dose adjustments will be assessed every 2 weeks from enrollment to 28 weeks gestation and then every 4 weeks from 29 weeks to delivery
  Mean number of LT4 dose adjustments needed according to etiology of hypothyroidism in each group
% of TSH values at goal according to anti-thyroid antibody status | TSH will be assessed every 2 weeks from enrollment to 28 weeks gestation and then every 4 weeks from 29 weeks to delivery
  TSH values within trimester specific goal range according to anti-thyroid antibody status

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Sullivan SD, Downs E, Popoveniuc G, Zeymo A, Jonklaas J, Burman KD. Randomized Trial Comparing Two Algorithms for Levothyroxine Dose Adjustment in Pregnant Women With Primary Hypothyroidism. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3499-3507. doi: 10.1210/jc.2017-01086. PMID 28911144